CLINICAL TRIAL: NCT01015027
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase 1 Study of the Safety and Tolerability of Intravenously Administered REGN668 in Healthy Volunteers
Brief Title: Ascending Dose Study of the Safety and Tolerability of REGN668(SAR231893) in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R668-AS-0907
Record Dates: First submitted 2009-11-10; First posted 2009-11-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 (Experimental): (3:1, active:placebo)
  Interventions: Biological: REGN668
- Dose 2 (Experimental): (3:1, active:placebo)
  Interventions: Biological: REGN668
- Dose 3 (Experimental): (3:1, active:placebo)
  Interventions: Biological: REGN668
- Dose 4 (Experimental): (3:1, active:placebo)
  Interventions: Biological: REGN668

INTERVENTIONS:
Biological: REGN668 — 4 IV Cohorts (Dose 1, 2, 3, & 4)

SUMMARY:
This study will test the safety and tolerability (how the body reacts to the drug) of REGN668 and placebo (an inactive substance that contains no medicine) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age.
2. Weight > 50 kg and < 120 kg.
3. For women of childbearing potential, a negative serum pregnancy test at the screening visit (visit 1) and a negative urine pregnancy test on day -1.
4. Willingness to refrain from the consumption of alcohol for 24 hours prior to each study visit.
5. For men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant) during the full duration of the study.
6. Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.
7. Able to read, understand and willing to sign the informed consent form.

Exclusion Criteria:

1. Onset of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to screening visit.
2. Pregnant or breast-feeding women.
3. Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that would adversely affect the subject's participation in this study.
4. Hospitalization for any reason within 60 days of screening (visit 1).
5. Known history of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C, and/or positive Hepatitis B surface antigen (HBsAg), positive Hepatitis C antibody (HCV).
6. Previous exposure to any therapeutic or investigational biological agent. results.
7. History of alcohol or substance abuse within previous 5 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in the study is the incidence of treatment-emergent adverse events in subjects treated with REGN668 or placebo, reported from the administration of study drug on day 1 to the completion of the study on day 85/visit 11. | 85 days

SECONDARY OUTCOMES:
Pharmacokinetics: Serum concentrations of REGN668 over time. | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Allen Radin, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Baltimore, Maryland, United States

REFERENCES:
- [Derived] Li Z, Radin A, Li M, Hamilton JD, Kajiwara M, Davis JD, Takahashi Y, Hasegawa S, Ming JE, DiCioccio AT, Li Y, Kovalenko P, Lu Q, Ortemann-Renon C, Ardeleanu M, Swanson BN. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Dupilumab in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2020 Aug;9(6):742-755. doi: 10.1002/cpdd.798. Epub 2020 Apr 29. PMID 32348036